CLINICAL TRIAL: NCT01170975
Title: An Open-label, Single-dose, Randomized, Crossover Study to Determine the Effects of Food on the Pharmacokinetics of Tesetaxel 10 mg Capsule in Solid Tumor Cancer Subjects
Brief Title: Effects of Food on the Pharmacokinetics of Tesetaxel 10 mg Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: TOPK103
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Solid Tumors
Keywords: Advanced solid tumors
MeSH Terms: interventions — tesetaxel; Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence 1 (Other): Treatment Period 1: Tesetaxel 10 mg in the fed state; Treatment Period 2: Tesetaxel 10 mg in the fasted state
  Interventions: Drug: Tesetaxel 10 mg with and then without food
- Treatment sequence 2 (Other): Treatment Period 1: Tesetaxel 10 mg in the fasted state; Treatment Period 2: Tesetaxel 10 mg in the fed state
  Interventions: Drug: Tesetaxel 10 mg without and then with food

INTERVENTIONS:
Drug: Tesetaxel 10 mg with and then without food — Treatment Period 1: Tesetaxel 10 mg in the fed state; Treatment Period 2: Tesetaxel 10 mg in the fasted state
  Arms: Treatment sequence 1
Drug: Tesetaxel 10 mg without and then with food — Treatment Period 1: Tesetaxel 10 mg in the fasted state; Treatment Period 2: Tesetaxel 10 mg in the fed state
  Arms: Treatment sequence 2

SUMMARY:
This study explores the effects of food (a high-fat meal) on the pharmacokinetics of tesetaxel.

DETAILED DESCRIPTION:
This study is being conducted to determine whether the pharmacokinetics of a single dose of tesetaxel administered as a capsule is affected by co-administration with food (a high-fat meal).

ELIGIBILITY:
Key inclusion criteria:

1. Male or female subjects between 18 and 75 years of age.
2. Histologically or cytologically confirmed advanced solid tumor malignancy.
3. Negative serum pregnancy test within 7 days prior to the first dose of study drug in women of childbearing potential.
4. Agreement to use a highly effective form of contraception throughout the treatment phase of the study in women of childbearing potential and sexually active men.
5. Body weight ≥ 50 kg for women and men and BMI within the range of 19 to 35 kg/m2 inclusive.
6. 12-lead ECG without any clinically significant abnormality as judged by the Investigator.
7. Able to swallow oral medication.
8. Adequate organ system function.

Key exclusion criteria:

1. A positive pre-study hepatitis B surface antigen.
2. Symptomatic or acute hepatic or biliary abnormalities.
3. Clinically significant gastrointestinal abnormalities that increase the risk for perforation.
4. Presence of uncontrolled infection.
5. Positive pre-study drug/alcohol screen.
6. Treatment with an investigational agent within the following time periods prior to the first dose of study drug: 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longest).
7. Current treatment with any cancer therapy that is causing significant gastrointestinal side effects, including but not limited to, nausea, vomiting, and diarrhea.
8. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with a subject's safety, obtaining informed consent, or compliance with the study.
9. Pregnancy or lactation.
10. Hypoalbuminemia (serum albumin <3.0 g/dL) at screening.
11. Consumption of red wine, seville oranges, grapefruit or grapefruit juice, and/or pummelos, exotic citrus fruits, or grapefruit hybrids within 14 days prior to the first dose of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | Predose and postdosing up to 36 days after administration of each dose
  Pharmacokinetic parameters include the area under the blood concentration-time curve (AUC0-inf, AUC0-t), concentration 24 h post dose (C24), maximum blood concentration (Cmax), time to maximum blood concentration (Tmax), terminal half-life (t½), and oral clearance (CL/F)

SECONDARY OUTCOMES:
Safety and tolerability | From screening through 36 days after administration of the final dose
  Adverse events, clinical laboratory tests, vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Harry W Alcorn, PharmD, Principal Investigator — Davita Clinical Research
Locations (1):
- DaVita Clinical Researh, Minneapolis, Minnesota, United States